CLINICAL TRIAL: NCT06670040
Title: Sham-Controlled rTMS for Refractory Depression in Autism Spectrum Disorder
Brief Title: Theta Burst Stimulation for Refractory Depression in Autism Spectrum Disorder
Acronym: RETSORE-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rana Elmaghraby, MD, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0682
Record Dates: First submitted 2024-10-16; First posted 2024-11-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ASD; Autism Spectrum Disorder; Autism; Depression - Major Depressive Disorder; MDD
Keywords: ASD; Autism; Autism Spectrum Disorder; MDD; Depression; TMS; TBS; Transcranial Magnetic Stimulation; Theta Burst Stimulation; Major Depressive Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Depression; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: It's a randomized controlled trial with active accelerated Theta Burst Stimulation (aTBS) treatment and sham controlled group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sham controlled (Sham Comparator): Sham aTBS targeting the left dorsolateral prefrontal cortex, 5 sessions per day for 5 days. If participants in the sham group do not show a significant treatment response by the 12-week follow-up - defined as a 50% reduction from baseline on the HDRS- they will then become eligible for and offered active, open-label treatment.
  Interventions: Procedure: Transcranial Magnetic Stimulation Sham
- Active TBS Treatment (Active Comparator): Active aTBS targeting the left dorsolateral prefrontal cortex, 5 sessions per day for 5 days.
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — All TBS sessions will be delivered at the same site, intensity (up to 90% RMT), pattern and duration. Treatment conditions differ only in the amount of intracranial activation induced (i.e., negligible activation in sham condition). TBS sessions consist of triplet 50 Hz bursts repeated every 200 msec (5 Hz), delivered to the left DLPFC in an intermittent (2 seconds on/8 seconds off) pattern for a total of 600 pulses per session; duration of 3 minutes 9 seconds.
  Arms: Active TBS Treatment
Procedure: Transcranial Magnetic Stimulation Sham — We will use a robust sham technique that suitably replicates the sensory experience (auditory and peripheral activation) of active TBS with minimal intracranial activation. The Magstim Horizon™ sham coil will be utilized for treatment delivery. This sham coil is visually identical to the active coil and replicates the sounds and sensation of the magnetic stimulation. All sham treatment will be delivered at the same site, intensity (up to 90% RMT), pattern and duration. Treatment conditions differ only in the amount of intracranial activation induced (i.e., negligible activation in sham condition). TBS sessions consist of triplet 50 Hz bursts repeated every 200 msec (5 Hz), delivered to the left DLPFC in an intermittent (2 seconds on/8 seconds off) pattern for a total of 600 pulses per session; duration of 3 minutes 9 seconds
  Arms: Sham controlled

SUMMARY:
Evaluate the efficacy of accelerated theta burst stimulation (aTBS) in reducing depressive symptoms in autism spectrum disorder (ASD)

DETAILED DESCRIPTION:
The overall goal of this study is to treat major depressive disorder (MDD) rapidly and effectively in individuals with autism spectrum disorder (ASD). Our central hypothesis is that accelerated theta burst stimulation (aTBS) targeting the left dorsal lateral prefrontal cortex (DLPFC) will significantly improve MDD symptoms and rate of remission compared to sham. We propose a double-blind RCT of 13-to 26-year-old individuals with ASD with MDD to test the efficacy of aTBS (n=12) versus sham (n=12) treatment. Participants will be rigorously characterized, including co-occurring conditions, any concurrent therapies, medications, social function, cognition, and sensory profile. A core battery of assessments will assess the efficacy of the intervention and maintenance of gains with respect to MDD and ASD-specific symptomology. Neural target engagement will be assessed by source-localized Electroencephalography (EEG) connectivity.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English and able to volunteer in the informed consent process and provide spontaneous narrative description of key elements, risks, and benefits of the study.
2. Aged 13-26, inclusive.
3. Full-scale intelligence quotient ≥ 70.
4. Diagnosis of ASD using criteria from Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Diagnosis will be confirmed by study psychologist/social worker and supported by scoring in the ASD on the Autism Diagnostic Observation Schedule (ADOS-2).
5. Diagnosis of MDD based on psychologist diagnosis and DSM-5-based structural diagnostic interview determine via KSADS
6. Exhibiting treatment resistance to at least one antidepressant drug treatment of adequate dose and duration.
7. Symptoms of moderate to severe depression according to Hamilton Depression Rating Scale ≥ 20 which must be maintained through lead-in period.
8. Participants are not required to discontinue current interventions but must agree to attempt to keep medications and other interventions stable during the study.

Exclusion Criteria:

1. Participation in an investigational drug trial within the past three months.
2. Active substance use disorder (excluding tobacco use) within the past 6 months.
3. Contraindications to Transcranial Magnetic Stimulation including, but not limited to, a history of epilepsy, the presence of metallic foreign bodies, or implanted medical devices (e.g. pacemaker, medical pump).
4. Actively suicidal (i.e., suicidal ideation with plan and intent) or deemed at high risk for suicide.
5. Current use of anticonvulsant, barbiturate, lithium, or benzodiazepine medications.
6. Prior rTMS treatment.
7. For female subjects of childbearing potential, a positive urine pregnancy test.

Ages: 13 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HDRS) | Completed at Screening, baseline, 2-week, 6-week, and 12-week follow up
  The HDRS is a 17-item rating scale administered by a trained rater following a semi-structured interview. Scores of 0-7 are generally within the normal range, and a score of 20 or higher indicates moderate depression severity. Research suggests that a decrement of 7 points on the HAMD-17 represents minimally clinically important differences from patient perspectives. HDRS will be assessed at screening, baseline and all follow up visits.
NIH Toolbox Cognition Battery | Completed at Screening, 2-week, 6-week, and 12-week follow up
  The NIH Toolbox was designed to serve as a brief, convenient set of measures to supplement other outcome measures in epidemiologic and longitudinal research and clinical trials.

SECONDARY OUTCOMES:
Electroencephalography (EEG) | Completed at baseline, 2-week, 6-week, and 12-week follow up
  Recordings are acquired using a gel-based electrode setup with a Biosemi EEG system, featuring 64 channels. Data are recorded at a sampling rate of 256 Hz, utilizing gel-based electrodes that enhance conductivity and minimize noise. This configuration ensures high-quality signal acquisition, enabling precise analysis of brain responses to various stimuli. EEG offers a real-time image of cortical excitability and connectivity. We will use power spectral analysis to assess changes in event-related gamma and alpha activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Elmaghraby, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All the IPD collected throughout this trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the completion of data collection